CLINICAL TRIAL: NCT01731938
Title: A Prospective, Single-blind, Randomized, Phase III Study to Evaluate the Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) as an Adjunct to Hemostasis During Soft Tissue Open Surgeries
Brief Title: Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) During Soft Tissue Open Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IG1103
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Soft Tissue Surgical Bleeding
Keywords: Fibrin Sealant; Soft tissue open surgery; Oxidized cellulose pads
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Sealant (FS) Grifols (Experimental): Fibrin Sealant Grifols consisting of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total).
  Interventions: Biological: Fibrin Sealant (FS) Grifols
- Surgicel® (Active Comparator): Surgicel® is a sterile, absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Interventions: Device: Surgicel®

INTERVENTIONS:
Biological: Fibrin Sealant (FS) Grifols — Fibrin Sealant (FS) Grifols: The maximum total volume of FS Grifols allowed to be applied at the target bleeding site by dripping or spraying was approximately 12 mL (equivalent to the full content of 2 FS Grifols kits).
  Arms: Fibrin Sealant (FS) Grifols
Device: Surgicel® — Up to four Surgicel® sheets applied to the target bleeding site according to Package Insert instructions and the surgeon's usual clinical practice.
  Other Names: Oxidized regenerated cellulose hemostat
  Arms: Surgicel®

SUMMARY:
This study is designed to assess the safety and efficacy of fibrin sealant (FS) Grifols in patients undergoing elective (non-emergency) soft tissue open surgery where bleeding may be present. The purpose of this study is to demonstrate that FS Grifols is not inferior to commercially-available oxidized cellulose pads (Surgicel®) in providing benefit in the time to hemostasis (i.e, the stoppage of bleeding). This study has a Preliminary Part (I) for study teams to become familiar with the application of FS Grifols and a Primary Part (II) to assess the safety and efficacy of FS Grifols. In both parts of the study, patients will be randomized in a 1:1 ratio to either FS Grifols or Surgicel.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin (Hgb) ≥ 8.0 g/dL at Baseline (within 24 hours prior to surgical procedure).
* Require elective (non-emergency), open (non-laparoscopic) surgical procedure involving soft (non-parenchymous) tissue.
* Target bleeding site is identified on soft tissue during urologic, gynecologic or general surgery procedures: 1) Simple or radical nephrectomies, 2) Total adrenalectomies, 3) Radical prostatectomies, 4) Pyeloplasties, 5) Radical cystectomies, 6) Simple or radical hysterectomies, 7) Lymphadenectomies (in the retroperitoneal or pelvic region only), 8) Retroperitoneal tumor resections, 9) Mastopexies, and 10) Abdominoplasties.
* A target bleeding site can be identified.
* Target bleeding site has moderate bleeding according to the Investigator's judgment.

Exclusion Criteria:

* Require thoracic, abdominal, retroperitoneal or pelvic surgery due to trauma.
* Infection in the anatomic surgical area.
* History of severe (e.g. anaphylactic) reactions to blood or to any blood-derived product.
* Previous known sensitivity to any FS Grifols component or any Surgicel® component.
* Females who are pregnant or nursing a child at Baseline (within 24 hours prior to surgical procedure).
* Receiving an organ transplant during the same surgical procedure.
* Undergone a therapeutic surgical procedure within 30 days from the screening visit.
* A target bleeding site cannot be identified.
* The target bleeding site has a mild or severe bleeding.
* Occurrence of major intraoperative complications that require resuscitation or deviation from the planned surgical procedure.
* Application of any topical haemostatic material on the cut soft tissue surface identified as the target bleeding site prior to application of the study treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (17):
  - 407, Florence, Alabama
  - 320, 322, 323, Pasadena, California
  - 404, Bridgeport, Connecticut
  - 321, Boynton Beach, Florida
  - 312, Rochester, Minnesota
  - 300, St Louis, Missouri
  - 327, Albany, New York
  - 305, New York, New York
  - 332, Poughkeepsie, New York
  - 304, Winston-Salem, North Carolina
  - 307, Pittsburgh, Pennsylvania
  - 325, Charleston, South Carolina
  - 331, Chattanooga, Tennessee
  - 314, Memphis, Tennessee
  - 402, Houston, Texas
  - 316, Houston, Texas
  - 405, Tacoma, Washington
- Hungary (5):
  - 702, Budapest
  - 701, Debrecen
  - 700, Debrecen
  - 703, Debrecen
  - 704, Győr
- Serbia (3):
  - 720, 722, 726, 723, Belgrade
  - 725, Niš
  - 721, 724, Novi Sad

RESULTS

PARTICIPANT FLOW:
Period: Preliminary Part I
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Started | 51 | 52
Completed | 48 | 44
Not Completed | 3 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Missed Week 6 visit | 0 | 3
Period: Primary Part II
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Started | 116 (Preliminary Part I was for study team familiarization with FS Grifols application.) | 108 (Subjects from Preliminary Part I were not carried over to Primary Part II to assess safety/efficacy.)
Completed | 103 | 95
Not Completed | 13 | 13
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 4 | 5
Not completed — Death | 2 | 1
Not completed — Missed Week 6 visit | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Fibrin Sealant (FS) Grifols Part I; Fibrin Sealant (FS) Grifols Part II: Fibrin Sealant Grifols consisting of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total).
  Fibrin Sealant (FS) Grifols: The maximum total volume of FS Grifols allowed to be applied at the target bleeding site by dripping or spraying was approximately 12 mL (equivalent to the full content of 2 FS Grifols kits).
- Surgicel® Part I; Surgicel® Part II: Surgicel® is a sterile, absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Surgicel®: Up to four Surgicel® sheets applied to the target bleeding site according to Package Insert instructions and the surgeon's usual clinical practice.
- Total: Total of all reporting groups
Arm/Group | Fibrin Sealant (FS) Grifols Part I | Surgicel® Part I | Fibrin Sealant (FS) Grifols Part II | Surgicel® Part II | Total
Number analyzed (Participants) | 51 | 52 | 116 | 108 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.17 (25.635) | 45.39 (25.024) | 48.51 (14.369) | 46.72 (14.330) | 47.21 (18.444)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 8 | 9 | 1 | 0 | 18
  Between 18 and 64 years | 27 | 28 | 98 | 90 | 243
  >=65 years | 16 | 15 | 17 | 18 | 66
Gender [Count of Participants; unit: Participants]
  Female | 27 | 28 | 87 | 86 | 228
  Male | 24 | 24 | 29 | 22 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 20 | 12 | 41
  Not Hispanic or Latino | 47 | 47 | 96 | 96 | 286
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1 | 2
  Black or African American | 5 | 5 | 22 | 25 | 57
  White | 46 | 46 | 93 | 81 | 266
  Not Specified | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Hemostasis Within 4 Minutes After Treatment Start
Description: Subjects achieving hemostasis at the target bleeding site within 4 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure.
Time Frame: From start of treatment until 4 minutes after treatment start
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Number analyzed (Participants) | 116 | 108
percentage of participants | 82.8 | 77.8

2. Secondary Outcome: Time to Hemostasis (TTH)
Description: TTH was measured from the start of treatment to the achievement of hemostasis at the target bleeding site, or to the end of the 10-minute observational period when hemostasis had not yet been achieved.
Time Frame: From start of treatment to the end of the 10-minute observational period
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Number analyzed (Participants) | 116 | 108
minutes | 3.6 (0.25) | 4.2 (0.29)

3. Secondary Outcome: Cumulative Proportion of Subjects Achieving Hemostasis at the Target Bleeding Site by 2 (T2), 3 (T3), 5 (T5), 7 (T7), and 10 (T10) Minutes After TStart.
Time Frame: From start of treatment to 2, 3, 5, 7, and 10 minutes after start of treatment
Measure: Number; unit: percentage of subjects
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Number analyzed (Participants) | 116 | 108
percentage of subjects
  Hemostasis by T2 | 53.4 | 43.5
  Hemostasis by T3 | 75.9 | 60.2
  Hemostasis by T5 | 83.6 | 78.7
  Hemostasis by T7 | 86.2 | 81.5
  Hemostasis by T10 | 89.7 | 83.3

4. Secondary Outcome: Treatments Failures
Description: The following were considered treatment failures:
  Persistent bleeding at the TBS beyond T4, Breakthrough (brisk and forceful) bleeding from the TBS that jeopardized subject safety according to the investigator's judgment at any moment during the 10 minute observational period and until TClosure, Re-bleeding at the TBS after the assessment of the primary efficacy endpoint at T4 and until TClosure Use of alternative hemostatic treatments or maneuvers (other than the study treatment) at the TBS during the 10-minute observational period and until TClosure or use of study treatment at the TBS beyond T4 and until TClosure.
Time Frame: From start of treatment to time of completion of surgical closure.
Measure: Number; unit: percentage of subjects
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Number analyzed (Participants) | 116 | 108
percentage of subjects | 17.2 | 22.2

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event data is based on the number of subjects who received study drug (safety population) in Preliminary Part (I) and Primary Part (II) of the study; 169 subjects in the FS Grifols group and 158 subjects in the Surgicel group. Two subjects who were randomized to the Surgicel treatment group received FS Grifols in error and are included in the FS Grifols treatment group.
Arm/Group | Fibrin Sealant (FS) Grifols | Surgicel®
Serious Adverse Events (participants affected / at risk) | 17/169 | 18/158
Other Adverse Events (participants affected / at risk) | 149/169 | 139/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrin Sealant (FS) Grifols (N=169) | Surgicel® (N=158)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrin Sealant (FS) Grifols (N=169) | Surgicel® (N=158)
Procedural pain (Injury, poisoning and procedural complications) | 92 (95) | 86 (86)
Procedural nausea (Injury, poisoning and procedural complications) | 24 (25) | 31 (31)
Nausea (Gastrointestinal disorders) | 23 (27) | 18 (19)
Constipation (Gastrointestinal disorders) | 19 (19) | 11 (11)
Pyrexia (General disorders) | 12 (12) | 15 (16)
Anemia (Blood and lymphatic system disorders) | 12 (12) | 14 (15)
Hypertension (Vascular disorders) | 13 (13) | 12 (12)
Vomiting (Gastrointestinal disorders) | 12 (13) | 9 (10)
Hypotension (Vascular disorders) | 11 (11) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10)
Incision site pain (Injury, poisoning and procedural complications) | 9 (9) | 7 (7)
Cervicitis (Infections and infestations) | 9 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing Sponsor at least thirty days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At Sponsor's request, the site will remove any confidential information (other than study results), and incorporate all reasonable comments by Sponsor, or delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor's Inventions.